CLINICAL TRIAL: NCT01070498
Title: Trichuris Suis Ova Therapy for Mild to Moderate Peanut and Tree Nut Allergy in Adults and Children
Brief Title: Trichuris Suis Ova in Peanut and Tree Nut Allergy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Food Allergy Initiative (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000414
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Food Allergy
Keywords: peanut hypersensitivity; tree nut hypersensitivity; allergy; Trichuris suis; hygiene hypothesis; treatment; clinical trial; food/adverse effect; peanut allergy (mild to moderate); tree nut allergy (mild to moderate)
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Nut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trichuris suis ova (TSO) (Experimental)
  Interventions: Drug: Trichuris suis ova (TSO)

INTERVENTIONS:
Drug: Trichuris suis ova (TSO) — Subjects will receive TSO every other week for 3 months. The dose will depend on the age of the subject and vary between 100 and 2500 eggs. TSO will be administered orally as a suspension in single dose vials prepared by Ovamed GmbH, a company not directly involved in the study.

SUMMARY:
The goal of this study is to determine whether Trichuris suis ova, a potential immunomodulator, is safe in adults and children allergic to peanut or tree nuts.

DETAILED DESCRIPTION:
Food allergy is a major cause of life-threatening hypersensitivity reactions. Currently avoidance of the allergenic food is the only established method of preventing reactions in allergic patients. This situation impacts significantly the lives of patients, mainly children, and their families. The current increase in the prevalence of allergic diseases, food allergy in particular, in the Western world has been attributed in part to changes in life style. Before the mid 20th century individuals were exposed to numerous bacterial, parasitic and viral agents. Since these times the progress of hygiene has considerably reduced the risk of exposure to these agents. It is thought that this lack of exposure, particularly during childhood, has led to subtle changes in humans' immune system resulting in an increased propensity to develop allergic and autoimmune responses, the so-called hygiene hypothesis. One of the means of reverting this propensity could be exposure to harmless biological agents. One such agent, eggs of the parasite Trichuris suis (Trichuris suis ova, TSO), has been shown to be well tolerated and efficient in patients with inflammatory bowel diseases. This phase I study will assess whether TSO is safe in adults and children with peanut or tree nut allergy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years old
* Positive skin-prick test to peanut or tree nut and a history of significant clinical symptoms within 60 minutes after the ingestion of peanuts or tree nuts.
* Peanut or tree nut allergy of mild to moderate grade based on the presence of localized or generalized erythema/urticaria/angioedema/oral pruritis, gastrointestinal symptoms, rhinoconjunctivitis, or mild laryngeal edema (voice change/tightening of throat/mild asthma), and the absence of symptoms/signs of severity (marked dyspnea, hypoxia, cyanosis, hypotension, confusion, incontinence, collapse or loss of consciousness)
* Otherwise in good health
* Ability to provide written informed consent

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise (cyanosis or SpO2 < 92% at any stage, confusion, collapse, loss of consciousness, or incontinence)
* Poor control of atopic dermatitis or current flare requiring an increase in atopic dermatitis medication
* Inability to discontinue antihistaminic for skin testing
* Severe persistent asthma as defined by the NHLBI criteria
* Asthma that requires oral steroids
* Asthma that has been controlled for less than 1 year
* FEV1<80% at the screening visit or immediately before the 1st administration of TSO
* Currently being treated with greater than medium daily doses of inhaled corticosteroids, as defined by the NHLBI guidelines
* Abnormal blood cell count
* Abnormal renal function (creatinine above twice the upper limit of normal range)
* Abnormal hepatic tests (AST, ALT above twice the upper limit of normal range)
* Allergy to Trichuris species
* Currently treated with anti-helminthic medication
* Previous treatment with immunosuppressive therapy, cytotoxic chemotherapy or lymphoid irradiation for any reason
* Insulin dependent diabetes
* History of HIV-1, HTLV-1 or Lyme disease
* Significant physical or mental disease that would preclude successful compliance and participation in the study, or, in the opinion of the investigators, constitute a hazard, such that enrollment in the study would not be in the subject's best interest
* Presence or history of cancer of any type except successfully treated basal cell or squamous cell carcinoma of the skin
* History of alcohol or drug abuse in the last 12 months; chronic liver or biliary disease
* Pregnancy and lactation; women of child bearing potential must have a documented negative pregnancy test at entry and at each visit during the study, and must be willing to practice adequate birth control during the duration of the study
* History of parasitism or positive stool determination for ova or parasite at screening
* Unwillingness or inability of patients (or caregivers) to give written consent or to follow the protocol successfully, including coming to the clinic every 2 weeks for about 4 months
* Currently participating in a study using an investigational new drug
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Presence in the household of an immunodeficient or immunosuppressed individual

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of unexpected severe side effects | every 2 weeks during the entire duration of the study
  Evidence of unexpected severe side effects due to the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Helene Jouvin, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States